CLINICAL TRIAL: NCT00177931
Title: Cefepime Pharmacokinetics in Liver Transplant Recipients in an Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: IRB # 0403014
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Evidence of Liver Transplantation
Keywords: Liver transplant; cefepime; antibiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers will be removed and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. All samples will be provided to investigators not associated with the study without any identifiers and only contain a code number. If a subject withdraws samples collected and not already processed will be destroyed.

GROUPS / COHORTS (1):
- liver transplant patients in ICU

SUMMARY:
The purposes of this study are to:

I. Characterize the plasma concentration-time profile of cefepime in liver transplant patients to determine the pharmacokinetic parameters in this patient population.

II. Perform stochastic modeling using the population pharmacokinetic parameters obtained in Specific Aim I to determine the ideal dose and dosing regimen of cefepime required to attain predetermined therapeutic targets in liver transplant patients.

DETAILED DESCRIPTION:
The use of cefepime in liver transplant patients at conventional doses used for other patient populations leads to non-optimal drug exposure among liver transplant patients. Furthermore, using serum creatinine as a method of estimating creatinine clearance is not the optimal way to determine the best cefepime dose. The consequence of this non-optimal exposure is the unattainability of therapeutic targets. These therapeutic targets are correlated with positive microbiologic outcome and clinical cure.

ELIGIBILITY:
Inclusion Criteria:

* Women and members of minority groups will be included in this study. However, as this study seeks to generate pilot data, there will be no specific statistical analysis comparing differences based on gender or race.
* Subjects receiving drugs known to induce or inhibit hepatic enzymes are not excluded from this study as cefepime is renally eliminated and not significantly metabolized by the liver.
* All liver transplant subjects are eligible for enrollment in this study, including subjects who have undergone a living related liver transplant.
* The pharmacokinetics of cefepime in children are significantly different from those of adults. For the purposes of this study only adults (aged > 18 years old) will be able to participate.

Exclusion Criteria:

* Subjects will be excluded if they are anemic (hemoglobin < 7 mg/dl), or are patients with severe gastrointestinal bleeding who are receiving packed red blood cells.
* Subjects who are receiving hemodialysis or other forms of renal replacement therapy (such as continuous veno-venous hemofiltration), or patients with a calculated creatinine clearance of < 10 ml/min will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patients in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2005-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
dead or alive post treatment | December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Brian Potoski, PharmD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States